CLINICAL TRIAL: NCT03841617
Title: The Use of 124-I-PET/CT Whole Body and Lesional Dosimetry in Differentiated Thyroid Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 190050; 19-DK-0050
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11-21

CONDITIONS: Thyroid Cancer
Keywords: Thyroid Cancer; PET/CT; 124-I; Radioiodine; Metastases
MeSH Terms: conditions — Thyroid Neoplasms; Neoplasm Metastasis | interventions — Thyrotropin Alfa; Iodine-131; Iodine-124

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 124I PET/CT scan after rhTSH (Active Comparator): 124I PET/CT scan after preparation with human recombinant TSH
  Interventions: Drug: Thyrogen; Radiation: I-131; Radiation: I-124
- 124I PET/CT scan after thyroid hormone withdrawal (Active Comparator): 124I PET/CT scan after preparation with thyroid hormone withdrawal
  Interventions: Radiation: I-131; Radiation: I-124; Other: Thyroid hormone withdrawal

INTERVENTIONS:
Drug: Thyrogen — intramuscular injection administered once/day for 2 consecutive days at Week 3; then once annually for subjects who meet criteria.
  Arms: 124I PET/CT scan after rhTSH
Radiation: I-131 — therapeutic dose administered orally to treat thyroid cancer at Week 8. 5-7 days later, the post-treatment I-131 Whole Body scan w/ SPECT is performed; then administered once annually, if the patient needs to be re-treated
Radiation: I-124 — one capsule ingested orally once at Week 3, and Week 8; then administered once annually to subjects who meet criteria.
Other: Thyroid hormone withdrawal — withdrawal of thyroid hormone during weeks 4 through 8
  Arms: 124I PET/CT scan after thyroid hormone withdrawal

SUMMARY:
Study rationale

High risk patients with differentiated thyroid cancer (DTC) require therapy with 131 I under thyroid stimulating hormone (TSH) stimulation. There are two methods of TSH stimulation endogenous by thyroid hormone withdrawal (THW) leading to hypothyroidism and exogenous by injection of human recombinant TSH (rhTSH Thyrogen). The appropriate 131-I activity utilized for treatment is either based on empiric fixed dosage choice or individually determined activity based on 131 I dosimetric calculations. Although dosimetry utilizing radioactive iodine isotope 131 I enables calculation of maximum safe dose, it does not estimate the tumoricidal activity necessary to destroy the metastatic lesions. The alternative radioactive isotope of iodine -124 I, used for positron emission tomography (PET) imaging, might be used for calculation not only the maximum safe131 I dose, but also to predict the absorbed dose in the metastatic lesions.

Study objectives

The primary objective of this study is to compare the 124 I -PET/CT lesional and whole body dosimetry in each individual patient with metastatic radioiodine (RAI)-avid thyroid cancer under preparation with rhTSH and THW. The secondary objective is to evaluate the predicted by PET/CT lesional uptake with the early response to therapy.

Study design

This is a phase 2 pilot prospective cohort study comparing the lesional and whole body dosimetry within each patient undergoing exogenous (rhTSH) and endogenous (THW) TSH stimulation and followed for 5 years.

Interventions

Each study participant will undergo rhTSH and THW-aided 124 I-PET/CT dosimetric evaluations and will be subsequently treated with THW-aided RAI activity based on dosimetric calculations enabling maximum safe dosage. The patients will be followed in 12+/-3 months intervals for 5 years.

Sample size and population

This pilot study will include 30 patients with high risk differentiated thyroid cancer presenting with distant and/or loco-regional metastases.

DETAILED DESCRIPTION:
Study Description:

Each study participant will undergo rhTSH and THW-aided 124IPET/ CT dosimetric evaluations and will be subsequently treated with THW-aided RAI activity based on dosimetric calculations enabling maximum safe dosage.

Objectives:

Primary objective: To compare the 124I -PET/CT lesional and whole body dosimetry in each individual patient with metastatic radioiodine (RAI)-avid thyroid cancer under preparation with rhTSH and THW.

Secondary objective: To evaluate the predicted by PET/CT lesional uptake with the early response to therapy.

Endpoints:

Primary Endpoint: The predicted radiation dose measured as rads per lesion compared per each measurable lesion between the dose calculated under rhTSH and under THW.

Secondary Endpoints: Area under the curve analyzing the association of dose per lesion measured in rads and objective response to treatment at 1, 2, 3, 4, 5 years landmarks.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients with established thyroid cancer diagnosis based on the pathology report reviewed at the National Institutes of Health, who:

  * underwent total thyroidectomy plus or minus neck lymph node dissection as clinically indicated,
  * are presenting with known per structural imaging (US neck, CT or MRI neck/chest/abdomen/pelvis) persistent/recurrent disease either locally advanced or presenting with distant metastases; or
  * are presenting with suspected persistent/recurrent locoregional or distant metastases based on the high risk features such as advanced tumor per pathology report (tumor size >4 cm, exrathyroidal extension, higher risk pathology such as tall cell, columnar cell, poorly differentiated variant, follicular thyroid cancer with gross vascular invasion, positive margins after the surgery, bulky lymphadenopathy in the central and/or lateral neck), detectable/increasing baseline/suppressed thyroglobulin (Tg) level or detectable/increasing anti-Tg antibody titers if anti-Tg antibodies are present.
  * are either RAI -naive or requiring repeated RAI therapy for locally advanced disease or distant metastases or underwent therapy with BRAF inhibitor (dabrafenib or vemurafenib*) or selumetinib** for at least 4 weeks that may re-induce RAI uptake.
  * Underwent imaging with either a CT or MRI of the brain and spine with gadolinium contrast to screen for the brain/spine metastases.

    * Age greater than or equal to 18 years of age.
    * 24 hour urine iodine excretion of less than or equal to 150 micro grams/24 hour.

      * BRAF inhibitors are recommended by 2021 NCCN guidelines as one of the management options for BRAF mutant tumors(13,14)

        * Selumetinib has an FDA orphan drug designation for adjuvant treatment of metastatic thyroid cancer to re-induce RAI uptake

EXCLUSION CRITERIA:

-Patients with RAI-non avid disease documented by negative post-therapy whole body scans performed after previous RAI treatments and not subjected to re-differentiation therapy.

* Serious underlying medical conditions that restrict diagnostic testing or therapy such as renal failure, congestive cardiac failure or active coexisting non-thyroid carcinoma, severe depression which might be exacerbated by thyroid hormone withdrawal.
* Patients with spinal or brain metastases as they are at risk of TSH-stimulation induced swelling of metastatic lesions leading to potentially detrimental side effects. These patients will be evaluated per the standard of care protocol 77-DK-0096.

  * Pregnant or lactating women per self report.
  * Adults who are incapable of providing informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2035-11-01 (Estimated); Study Completion 2035-11-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the whole body and lesional 124I uptake within each patient prepared for imaging with human recombinant TSH (rhTSH) and thyroid hormone withdrawal (THW) | 9 weeks
  Whole body and lesional uptake of 124I calculated after preparation with human recombinant TSH (rhTSH) compared to dosimetry calculated after preparation using thyroid hormone withdrawal (THW)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Klubo-Gwiezdzinska, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Subject level data will be shared upon request after appropriate collaboration agreements are in place.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-DK-0050.html